CLINICAL TRIAL: NCT03221452
Title: Adaptation of a Cognitive Training Intervention for Diabetes Self-Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-08-0001
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Cognitive Function Abnormal; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Cognition Disorders; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Single group study for intervention feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): The intervention includes 4 every other week, 2-hour educational sessions to teach compensatory strategies along with skill development and training. Educational sessions will include content on common cognitive problems experienced by people with T2DM and discussion of compensatory strategies to improve cognitive skills as well as content on behaviors and lifestyle strategies to maintain cognitive functioning. Each participant will use the online training program (BrainHQ/Posit Science) for a minimum of 45 minutes 3 times a week and to record practice times and dates. Tasks in the computer training are arranged so that as the user moves forward, the tasks become more challenging. Each task is in a game-like format.
  Interventions: Behavioral: Memory, Attention, and Problem Solving Skills for Diabetes

INTERVENTIONS:
Behavioral: Memory, Attention, and Problem Solving Skills for Diabetes — Classes will include: (1) information on diabetes self-management including glucose self-monitoring and medication management; (2) assessment of cognitive problems; (3) resources and barriers to self-management; and (4) lifestyle changes to maximize cognitive health. Participants will also practice those skills with online computer games.

SUMMARY:
The aims of this project are: (1) to refine an existing cognitive rehabilitation intervention and tailor it for persons with T2DM by using current literature and interview data from 10 participants with T2DM and (2) to conduct a feasibility study of the adapted intervention with 20 participants with T2DM. The intervention consists of 8 weekly group educational sessions to teach compensatory cognitive strategies. Participants will also use a web-based, game-like program to build on the didactic information and practice activities to improve cognitive health.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) increases the risk for cognitive impairment and doubles the rate of cognitive decline after diabetes is diagnosed. In turn, the presence of cognitive dysfunction can make diabetes self-management more difficult. Few interventions have attempted to focus on cognitive function in the context of diabetes and none, to date have tested an intervention to improve cognition in order to improve diabetes self-management. Therefore the aims of this project are: (1) to refine an existing cognitive rehabilitation intervention and tailor it for persons with T2DM by using current literature and interview data from 10 participants with T2DM and (2) to conduct a feasibility study of the adapted intervention with 20 participants with T2DM. The intervention consists of 8 weekly group educational sessions to teach compensatory cognitive strategies. Additionally, participants will use a web-based, game-like program to build on the didactic information and practice activities to improve cognitive health. The project will provide baseline data for further research on diabetes self-management in the context of cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 70
* Have been diagnosed with type 2 diabetes for at least 2 years
* Score of at least 10 on the Perceived Deficits Questionnaire
* Read and write in English
* Have access to transportation and telephone and Internet services

Exclusion Criteria:

* limitations that preclude study activities
* have been diagnosed with dementia or disorders that can affect cognition such as depression
* type 1 diabetes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetes Self-Care Activities | Baseline and immediately post-intervention
  Summary of Diabetes Self-Care Activities Questionnaire; 18 items; Participants answer questions regarding how many days in the last week have they performed a certain aspect of diabetes self-management behaviors such as diet, smoking, and physical activity.

SECONDARY OUTCOMES:
General Self-Efficacy Scale | Baseline and immediately post-intervention
  10 items; confidence in ability to influence outcomes. Responses are made on a 4-point scale (1 = not true at all, 2= hardly true, 3 = moderately true, 4= exactly true) to items such as "I can always manage to solve difficult problems If I try hard enough."
Multifactorial Memory Questionnaire | Baseline and immediately post-intervention
  57 items; assesses contentment with one's memory, subjective memory capability, and use of memory aids. Participants rate their level of agreement with each item on a 5-point scale (strongly agree = 1, agree = 2, undecided = 3, disagree = 4, strongly disagree = 5) for the Contentment subscale; The Ability subscale asks participants to indicate the frequency with which each memory failure has occurred in the past 2 weeks on a 5-point scale (all the time = 1, often =2, sometimes = 3, rarely =4, never =5); The third subscale, Strategy, asks participants to rate the frequency of use of certain memory strategies on a 5-point scale (never =1, rarely =2, sometimes =3, often =4, all the time =5).
Change in executive function | Baseline and immediately post-intervention
  Barkley Deficits in Executive Functioning Scale - Short Form Scale; 20 items assessing the frequency at which participants have exhibited certain behaviors in specific executive functioning areas over the past 6 months. The areas include: self-management to time, self-organization/problem-solving, self-restraint, self-motivation, and self-regulation of emotion. Items are measured using a 4-point Likert scale, ranging from never or rarely (1) to very often (4).
Center for Epidemiologic Studies Depression Scale | Baseline and immediately post-intervention
  20 items; measurement of depressive symptoms. Participants indicate responses on a 4-point item scale from rarely/none of the time to most/all of the time in 8 health dimensions: role limitations due to physical problems, social functioning, physical functioning, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Heather E Cuevas, PhD, Principal Investigator — The University of Texas at Austin

IPD SHARING:
Plan to Share IPD: No